CLINICAL TRIAL: NCT04484883
Title: Performance of Six Equations for Estimating Resting Energy Expenditure in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 6/2020
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observational
  Other Names: Retrospective cohort study

SUMMARY:
The present study evaluated the statistical and clinical performance of the six common equations in subjects with type 2 diabetes adopting indirect calorimetry as reference standard

DETAILED DESCRIPTION:
All consecutive subjects with type 2 diabetes referred from June 2012 to December 2019 were eligible. They were excluded if data on ongoing therapy, anthropometric or laboratory parameters, or measured REE was not available or if presenting with conditions known to affect indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Available resting energy expenditure assessed by indirect calorimetry

Exclusion Criteria:

* data on ongoing therapy (e.g. lifestyle measures with or without approved drugs), anthropometric or laboratory parameters (including white blood count, estimated glomerular filtration rate, TSH), or REE assessed by the means of indirect calorimetry could not be retrieved
* presenting with conditions known to affect indirect calorimetry (e.g. patients with strenuous exercise on the day before, asymptomatic patients with severe chronic kidney disease (eGFR < 30 ml/min/ 1.73 m2), increased white blood count, or subnormal TSH)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 250 patients (124 females and 126 males, mean age 61.9 ± 8.5 years)
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline
  Body weight in Kilograms
Neck circumference | Baseline
  Neck circumference in cm
Waist circumference | At baseline
  Waist circumference in cm
Hip circumference | Baseline
  Hip circumference in cm
Body mass index (BMI) | At baseline
  Body mass index (BMI) (expressed in kg/m^2)
Resting Energy Expenditure (REE) | At baseline
  Resting Energy Expenditure (REE) in kcal

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Gastroenterology IRCCS S. de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No